CLINICAL TRIAL: NCT06273878
Title: From Fetal-maternal Interface Immune Tolerance to Endometrial Cancer Immune Escape: Potential Targets for Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Sponsor
Other Study IDs: RS1439/20
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-interventional retro-prospective study on Endometrial tissue samples taken from surgically treated patients.

DETAILED DESCRIPTION:
The picture of precisely coordinated immune adaptations over time at the maternal-fetal interface level and altered in pregnancy complications, could reveal a specific "immune clock" in tumors. The study aims to decipher mechanisms of immunodeficiency by helping to predict recurrence in patients with endometrial cancer and identify molecular pathways that are turned on or off in progression from lesions early to advanced neoplasia. This will allow the discovery of potential immunotherapy targets to interfere with the immune escape activation process or to reactivate/re-educate the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Histological diagnosis of endometrial hyperplasia with and without atypia, carcinoma of the endometrium histotype endometrioid at any stage of the disease (FIGO I-IV), patients subjected to hysterectomy for benign extra-endometrial pathology, patients with recurrence/metastasis from endometrioid endometrial carcinoma that are subjected to surgery;
* Adequate biological material to be able to carry out the analyzes previously described;
* Written informed consent (only for patients in the prospective part and/or in follow-up);
* For the retrospective part: availability of samples adequately stored at the Institute biobank and availability of follow-up data.

Exclusion Criteria:

* Comorbidities not controlled with adequate medical therapy;
* Infections of the endometrial cavity (pyometra);
* Synchronous tumors;
* Neoadjuvant treatments;
* Previous radiation treatments on the pelvic region.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The population is represented by patients with endometrial cancer who have undergone, or who have will undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Validate the differential expression of LOX-1 and NALP3 receptors. | 36 months
  Validate the differential expression of LOX-1 and NALP3 receptors at different steps progression of endometrial cancer; identify immune signatures shared between using transcriptomics the maternal-fetal interface and the different stages of progression of endometrial cancer; investigate their role functional in the immune escape process in endometrial carcinoma and/or in the pro-inflammatory response.

SECONDARY OUTCOMES:
Characterize phenotypic alterations. | 36 months
  Characterize the phenotype and functional alterations of multiple candidate biomarkers relevant selected in AIM1 (surface antigens / cytokines / molecular pathways), a level of the cells of the immune infiltrate, in the different stages of cancer progression to the endometrium.
Evaluate the predictive and/or prognostic value. | 36 months
  Evaluate the predictive and/or prognostic value of the immuno-score deriving from the data of Aim 1 and Aim 2 alone or in combination with clinical and prognostic risk factors known histopathological findings, expressed in the ESMO-ESGO-ESTRO consensus conference.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - National Cancer Institute - IFO -, Rome, RM
  - "Regina Elena" National Cancer Institute, Rome